CLINICAL TRIAL: NCT03011892
Title: A Phase 2, Randomized, Dose-Ranging, Vehicle-Controlled and Triamcinolone 0.1% Cream-Controlled Study to Evaluate the Safety and Efficacy of INCB018424 Phosphate Cream Applied Topically to Adults With Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Ruxolitinib Phosphate Cream Applied Topically to Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-206
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; eczema; pruritus; Janus kinase (JAK) inhibitors
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus | interventions — ruxolitinib; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Double Blind (DB): Vehicle BID (Placebo Comparator): Participants applied vehicle cream twice daily (BID) for 8 weeks DB period.
  Interventions: Drug: Vehicle Cream BID
- DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID (Active Comparator): Participants applied triamcinolone 0.1% cream BID for 4 weeks followed by vehicle cream for 4 weeks in DB period.
  Interventions: Drug: Triamcinolone 0.1% Cream BID; Drug: Vehicle Cream BID
- DB: Ruxolitinib 0.15% Once Daily (QD) (Experimental): Participants applied ruxolitinib 0.15% cream QD for 8 weeks in DB period.
  Interventions: Drug: Ruxolitinib 0.15% Cream QD
- DB: Ruxolitinib 0.5% QD (Experimental): Participants applied ruxolitinib 0.5% cream QD for 8 weeks in DB period.
  Interventions: Drug: Ruxolitinib 0.5% Cream QD
- DB: Ruxolitinib 1.5% QD (Experimental): Participants applied ruxolitinib 1.5% cream QD for 8 weeks in DB period.
  Interventions: Drug: Ruxolitinib 1.5% Cream QD
- DB: Ruxolitinib 1.5% BID (Experimental): Participants applied ruxolitinib 1.5% cream BID for 8 weeks in DB period.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- Open-Label (OL): Vehicle BID to Ruxolitinib 1.5% BID (Placebo Comparator): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- OL: TAC BID/Vehicle BID to Ruxolitinib 1.5% BID (Active Comparator): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID (Experimental): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID (Experimental): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID (Experimental): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID
- OL: Ruxolitinib 1.5% BID to Ruxolitinib 1.5% BID (Experimental): Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
  Interventions: Drug: Ruxolitinib 1.5% Cream BID

INTERVENTIONS:
Drug: Ruxolitinib 0.15% Cream QD — Ruxolitinib 0.15% cream QD
  Other Names: INCB018424
  Arms: DB: Ruxolitinib 0.15% Once Daily (QD)
Drug: Ruxolitinib 0.5% Cream QD — Ruxolitinib 0.5% cream QD
  Other Names: INCB018424
  Arms: DB: Ruxolitinib 0.5% QD
Drug: Ruxolitinib 1.5% Cream QD — Ruxolitinib 1.5% cream QD
  Other Names: INCB018424
  Arms: DB: Ruxolitinib 1.5% QD
Drug: Ruxolitinib 1.5% Cream BID — Ruxolitinib 1.5% cream BID
  Other Names: INCB018424
  Arms: DB: Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% BID to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID; OL: TAC BID/Vehicle BID to Ruxolitinib 1.5% BID; Open-Label (OL): Vehicle BID to Ruxolitinib 1.5% BID
Drug: Triamcinolone 0.1% Cream BID — Triamcinolone 0.1% cream BID
  Arms: DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID
Drug: Vehicle Cream BID — Vehicle cream BID
  Arms: DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID; Double Blind (DB): Vehicle BID

SUMMARY:
The purpose of this study is to establish the efficacy of each strength of ruxolitinib cream once daily (QD) or twice daily (BID) in participants with atopic dermatitis as compared with vehicle cream BID.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with atopic dermatitis (AD) as defined by the Hanifin and Rajka criteria.
* Participants with a history of AD for at least 2 years.
* Participants with an Investigator's Global Assessment (IGA) score of 2 to 3 at screening and baseline.
* Participants with body surface area (BSA) of AD involvement, excluding the face and intertriginous areas, of 3% to 20% at screening and baseline.
* Participants who agree to discontinue all agents used to treat AD from screening through the final follow-up visit.

Exclusion Criteria:

* Participants with evidence of active acute or chronic infections.
* Use of topical treatments for AD (other than bland emollients) within 2 weeks of baseline.
* Systemic immunosuppressive or immunomodulating drugs (eg, oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolate mofetil, azathioprine) within 4 weeks or 5 half-lives of baseline (whichever is longer).
* Participants with other dermatologic disease besides AD whose presence or treatments could complicate the assessment of disease (eg, psoriasis).
* Participants with a history of other diseases besides dermatologic disorders (eg, other autoimmune diseases) taking treatments that could complicate assessments.
* Participants with cytopenias at screening, defined as:

  * Leukocytes < 3.0 × 10^9/L.
  * Neutrophils < lower limit of normal.
  * Hemoglobin < 10 g/dL.
  * Lymphocytes < 0.8 × 10^9/L
  * Platelets < 100 × 10^9/L.
* Participants with severely impaired liver function (Child-Pugh Class C) or end-stage renal disease (ESRD) on dialysis or at least 1 of the following:

  * Serum creatinine > 1.5 mg/dL.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 × upper limit of normal.
* Participants taking potent systemic cytochrome P450 3A4 inhibitors or fluconazole within 2 weeks or 5 half-lives, whichever is longer, before the baseline visit (topical agents with limited systemic availability are permitted).
* Participants who have previously received Janus kinase (JAK) inhibitors, systemic or topical (e.g., ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD, Study Director — Incyte Corporation
Locations (52):
- United States (35):
  - UAB DERMATOLOGY, 2000 6th Avenue South, Birmingham, Alabama
  - BURKE PHARMACEUTICAL RESEARCH, 601 W. Commerce, Bryant, Arkansas
  - ENCINO RESEARCH CENTER, 16133 Ventura Blvd, Encino, California
  - DERMATOLOGY RESEARCH ASSOCIATES,8930 South Sepulveda Blvd, Los Angeles, California
  - DERMATOLOGY SPECIALISTS, INC, 3629 Vista Way, Oceanside, California
  - INTEGRATED RESEARCH GROUP, INC, 4646 Brockton Avenue, Riverside, California
  - SAN LUIS DERMATOLOGY AND LASER CLINIC, 15 Santa Rosa Street, San Luis Obispo, California
  - NEW ENGLAND RESEARCH ASSOCIATES LLC, 5520 Park Avenue, Trumbull, Connecticut
  - DS RESEARCH, 2241 Green Valley Road, New Albany, Indiana
  - THE INDIANA CLINICAL TRIALS CENTER, 824 Edwards Drive, Plainfield, Indiana
  - DERMRESEARCH, 1169 Eastern Parkway 2310, Louisville, Kentucky
  - DS RESEARCH, 3810 Springhurst Blvd, Louisville, Kentucky
  - ACTIVMED PRACTICES & RESEARCH, INC, 138 Conant Street, Beverly, Massachusetts
  - TUFTS MEDICAL CENTER, 800 Washington Street, Boston, Massachusetts
  - HENRY FORD HOSPITAL, 3031 West Grand Blvd, Detroit, Michigan
  - WASHINGTON UNIVERSITY - DERMATOLOGY, 4921 Parkview Place, St Louis, Missouri
  - WASHINGTON UNIVERSITY - DERMATOLOGY, 969 Mason Road, St Louis, Missouri
  - ACTIVMED PRACTICES AND RESEARCH, INC, 110 Corporate Drive, Portsmouth, New Hampshire
  - HASSMAN RESEARCH INSTITUTE, LLC, 175 Cross Keys Road, Berlin, New Jersey
  - DERMATOLOGY CONSULTING SERVICES, PLLC, 2444 North Main Street, High Point, North Carolina
  - WAKE RESEARCH ASSOCIATES LLC, 3100 Duraleigh Road, Raleigh, North Carolina
  - DERMATOLOGISTS OF GREATER COLUMBUS, 2359 East Main Street, Bexley, Ohio
  - RAPID MEDICAL RESEARCH, INC, 3619 Park East Drive, Cleveland, Ohio
  - CENTRAL SOONER RESEARCH, 900 North Porter, Norman, Oklahoma
  - PARISH DERMATOLOGY, INC, 1845 Walnut Street, Philadelphia, Pennsylvania
  - PEAK RESEARCH LLC, 2589 Washington Rd, Upper Saint Clair, Pennsylvania
  - ARLINGTON RESEARCH CENTER, INC, 711 East Lamar Blvd, Arlington, Texas
  - DERMRESEARCH INC., 8140 North Mopac Expressway, Austin, Texas
  - J&S STUDIES, INC, 1710 Crescent Pointe Pkwy, College Station, Texas
  - CENTER FOR CLINICAL STUDIES (CCS), 1401 Binz, Houston, Texas
  - SUZANNE BRUCE AND ASSOCIATES, PA, 1900 St. James Place, Houston, Texas
  - CLINICAL TRIALS OF TEXAS, INC, 7940 Floyd Curl Drive, San Antonio, Texas
  - DERMATOLOGY CLINICAL RESEARCH CENTER OF SAN ANTONIO, 7810 Louis Pasteur, San Antonio, Texas
  - CENTER FOR CLINICAL STUDIES, 451 North Texas Avenue, Webster, Texas
  - CHARLOTTESVILLE DERMATOLOGY, 600 Peter Jefferson Parkway, Charlottesville, Virginia
- Canada (17):
  - INSTITUTE FOR SKIN ADVANCEMENT, 4935 40th Avenue Nw, Calgary, Alberta
  - DR. CHIH-HO HONG MEDICAL INC., 15300 105 Avenue, Surrey, British Columbia
  - WISEMAN DERMATOLOGY RESEARCH INC, 6 - 1170 Taylor Avenue, Winnipeg, Manitoba
  - CCA MEDICAL RESEARCH, 95 Bayly Street West, Ajax, Ontario
  - SIMCODERM MEDICAL AND SURGICAL DERMATOLOGY CENTER, 5 Quarry Ridge Road, Barrie, Ontario
  - LYNDERM RESEARCH INC, 25 Main Street Markham North, Markham, Ontario
  - DERMEDGE RESEARCH INC., 333 Lakeshore Road West, Mississauga, Ontario
  - NORTH BAY DERMATOLOGY CENTRE, 500 Cassells Street, North Bay, Ontario
  - RESEARCH BY ICLS, 1344 Cornwall Road, Oakville, Ontario
  - OFFICE OF DR. MICHAEL ROBERN, 1 Centrepointe Drive, Ottawa, Ontario
  - SKIN CENTRE FOR DERMATOLOGY, 775 Monaghan Road, Peterborough, Ontario
  - YORK DERMATOLOGY CENTER, 250 Harding Blvd West, Richmond Hill, Ontario
  - RESEARCH TORONTO, 208 Bloor Street West, Toronto, Ontario
  - K. PAPP CLINICAL RESEARCH, 135 Union Street East, Waterloo, Ontario
  - XLR8 MEDICAL RESEARCH, 2425 Tecumseh Road East, Windsor, Ontario
  - WINDSOR CLINICAL RESEARCH INC, 2224 Walker Road, Windsor, Ontario
  - CLINIQUE DERMATOLOGIQUE DE SAINT-JEROME, 555 Boul. Saint-antoine, Saint-Jérôme, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong X, Chen X, Kuligowski ME, Liu X, Liu X, Cimino E, McGee R, Yeleswaram S. Pharmacokinetics of Ruxolitinib in Patients with Atopic Dermatitis Treated With Ruxolitinib Cream: Data from Phase II and III Studies. Am J Clin Dermatol. 2021 Jul;22(4):555-566. doi: 10.1007/s40257-021-00610-x. Epub 2021 May 12. PMID 33982267
- [Derived] Kim BS, Howell MD, Sun K, Papp K, Nasir A, Kuligowski ME; INCB 18424-206 Study Investigators. Treatment of atopic dermatitis with ruxolitinib cream (JAK1/JAK2 inhibitor) or triamcinolone cream. J Allergy Clin Immunol. 2020 Feb;145(2):572-582. doi: 10.1016/j.jaci.2019.08.042. Epub 2019 Oct 17. PMID 31629805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 307 participants were randomized and 306 were treated at 50 study centers in the United States and Canada from 9 January 2017 to 12 March 2018.
Pre-assignment Details: 307 participants randomized to 6 treatment groups (ruxolitinib cream 1.5% BID, or QD, 0.5% or 0.15% QD, vehicle BID, & TAC 0.1% BID). Participants applied blinded study drug for 8 weeks, TAC 0.1% BID for 4 weeks followed by vehicle BID for 4 weeks in DB period. After DB period, participants who met criteria (compliant with the protocol and no safety concerns) offered OL treatment with ruxolitinib 1.5% BID for 4 weeks. Out of 261 participants who completed DB Period, 252 entered the OL Period.
Groups:
- OL: TAC BID/ Vehicle BID to Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% Cream BID for 8 Weeks in DB Period.: Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
Period: Double Blind (DB) Period
Arm/Group | Double Blind (DB): Vehicle BID | DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% Once Daily (QD) | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID | Open-Label (OL): Vehicle BID to Ruxolitinib 1.5% BID | OL: TAC BID/ Vehicle BID to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% Cream BID for 8 Weeks in DB Period.
Started | 52 | 51 | 51 | 51 | 52 | 50 | 0 | 0 | 0 | 0 | 0 | 0
Treated in DB Period (One participant was randomized but did not receive study drug.) | 52 | 51 | 51 | 51 | 51 | 50 | 0 | 0 | 0 | 0 | 0 | 0
Completed Treatment Through Week 4 | 44 | 46 | 48 | 47 | 49 | 49 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed= Number of participants who completed treatment through Week 8 in DB period.) | 41 | 41 | 45 | 44 | 45 | 45 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 10 | 6 | 7 | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 1 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label (OL) Period
Arm/Group | Double Blind (DB): Vehicle BID | DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% Once Daily (QD) | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID | Open-Label (OL): Vehicle BID to Ruxolitinib 1.5% BID | OL: TAC BID/ Vehicle BID to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% Cream BID for 8 Weeks in DB Period.
Started | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 40 | 45 | 41 | 42 | 43
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 37 | 43 | 41 | 40 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 2 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 2
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who are randomized to the study.
Groups:
- DB : Ruxolitinib 0.5% QD: Participants applied ruxolitinib 0.5% cream QD for 8 weeks in DB period.
- DB : Ruxolitinib 1.5% QD: Participants applied ruxolitinib 1.5% cream QD for 8 weeks in DB period.
- DB : Ruxolitinib 1.5% Cream Twice Daily (BID): Participants applied ruxolitinib 1.5% cream BID for 8 weeks in DB period.
- Total: Total of all reporting groups
Arm/Group | Double Blind (DB): Vehicle BID | DB: Triamcinolone (TAC) 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% Once Daily (QD) | DB : Ruxolitinib 0.5% QD | DB : Ruxolitinib 1.5% QD | DB : Ruxolitinib 1.5% Cream Twice Daily (BID) | Total
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 52 | 50 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (15.04) | 38.5 (16.19) | 38.4 (13.83) | 38.6 (13.73) | 39.1 (14.54) | 39.0 (15.72) | 38.1 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 26 | 27 | 31 | 24 | 168
  Male | 20 | 23 | 25 | 24 | 21 | 26 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 2 | 3 | 1 | 3 | 20
  Not Hispanic or Latino | 47 | 43 | 49 | 48 | 51 | 47 | 285
  Other | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 27 | 28 | 27 | 33 | 24 | 33 | 172
  Black/African-American | 15 | 13 | 17 | 10 | 17 | 13 | 85
  Asian | 8 | 8 | 5 | 8 | 10 | 2 | 41
  Native Hawaiian/Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 2 | 2 | 0 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 4 in Participants Treated With Ruxolitinib 1.5% Cream Twice a Day (BID) Compared With Participants Treated With Vehicle Cream BID
Description: EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 areas of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Time Frame: Baseline and Week 4
Population: Participants from Intent to treat (ITT) population, all participants who are randomized to vehicle BID or ruxolitinib 1.5% BID, with available data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- DB: Vehicle BID: Participants applied vehicle cream BID for 8 weeks in DB period.
Arm/Group | DB: Vehicle BID | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 44 | 49
percent change | -11.90 (6.65) | -71.57 (6.42)
Statistical Analysis 1: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% BID; Test type: Superiority; p < 0.0001, MMRM; Difference in Least Square (LS) Mean = -59.66, 95% CI 2-sided [-77.85 to -41.47]

2. Secondary Outcome: Mean Percentage Change From Baseline in EASI Score at Week 4 in Participants Treated With Ruxolitinib QD Compared With Participants Treated With Vehicle Cream BID
Description: as for outcome 1
Time Frame: Baseline and Week 4
Population: Participants from Intent to treat (ITT) population, all participants who are randomized to vehicle BID and ruxolitinib 0.15% or 0.5% or 1.5% QD in the DB Period, with available data were included in the analysis
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- DB: Ruxolitinib 0.15% QD: Participants applied ruxolitinib 0.15% cream QD for 8 weeks in DB period.
Arm/Group | DB: Vehicle BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD
Number analyzed (Participants) | 44 | 47 | 47 | 49
percent change | -11.90 (6.65) | -44.92 (6.47) | -52.80 (6.52) | -66.72 (6.36)
Statistical Analysis 1: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.15% QD; DB: Vehicle BID, Ruxolitinib 0.15% QD; Test type: Superiority; p = 0.0004, MMRM; Difference in LS Mean = -33.01, 95% CI 2-sided [-51.27 to -14.76]
Statistical Analysis 2: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.5% QD; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -40.90, 95% CI 2-sided [-59.23 to -22.57]
Statistical Analysis 3: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% QD; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -54.82, 95% CI 2-sided [-72.93 to -36.70]

3. Secondary Outcome: Mean Percentage Change From Baseline in EASI Score at Week 4 in Participants Treated With Ruxolitinib QD/BID Cream Compared With Participants Treated With Triamcinolone 0.1% Cream BID Followed by Vehicle
Description: as for outcome 1
Time Frame: Baseline and Week 4
Population: Participants from ITT population, all participants who are randomized to TAC 0.1% BID followed by vehicle BID and ruxolitinib 0.15% or 0.5% or 1.5% QD/BID in the DB Period, with available data were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- DB: TAC 0.1% BID/Vehicle Cream BID: Participants applied triamcinolone 0.1% cream BID for 4 weeks followed by vehicle cream for 4 weeks in DB period.
Arm/Group | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 46 | 47 | 47 | 49 | 49
percent change | -59.54 (6.53) | -44.92 (6.47) | -52.80 (6.52) | -66.72 (6.36) | -71.57 (6.42)
Statistical Analysis 1: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.15% QD; Triamcinolone 0.1% BID/Vehicle Cream BID, DB: Ruxolitinib 0.15% QD; Test type: Superiority; p = 0.1127, MMRM; Difference in LS Mean = 14.63, 95% CI 2-sided [-3.47 to 32.73]
Statistical Analysis 2: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.5% QD; Triamcinolone 0.1% BID/Vehicle Cream BID, DB: Ruxolitinib 0.5% QD; Test type: Superiority; p = 0.4659, MMRM; Difference in LS Mean = 6.74, 95% CI 2-sided [-11.44 to 24.92]
Statistical Analysis 3: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% QD; Triamcinolone 0.1% BID/Vehicle Cream BID, DB: Ruxolitinib 1.5% QD; Test type: Superiority; p = 0.4320, MMRM; Difference in LS Mean = -7.18, 95% CI 2-sided [-25.13 to 10.77]
Statistical Analysis 4: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% BID; Test type: Superiority; p = 0.1903, MMRM; Difference in LS Mean = -12.02, 95% CI 2-sided [-30.05 to 6.00]

4. Secondary Outcome: Mean Percentage Change From Baseline in EASI Score at Week 2 and Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 2 and 8
Population: ITT Population included all participants who are randomized to Vehicle BID, TAC 0.1% BID/Vehicle Cream BID, Ruxolitinib 0.15%, 0.5%, 1.5%, 1.5% QD/BID in the DB Period. The overall number of participants analyzed are participants with data available for analysis for this Outcome Measure and "n" signifies number of participants with data available at specific timepoint.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 52 | 50
percent change
  Week 2: number analyzed (Participants) | 48 | 49 | 50 | 46 | 51 | 49
  Week 2 | -4.84 (5.34) | -39.94 (5.29) | -29.96 (5.23) | -45.88 (5.41) | -49.88 (5.18) | -52.68 (5.29)
  Week 8: number analyzed (Participants) | 41 | 43 | 45 | 43 | 46 | 44
  Week 8 | -21.86 (7.09) | -58.02 (6.94) | -50.24 (6.82) | -58.37 (6.93) | -67.05 (6.72) | -79.01 (6.83)
Statistical Analysis 1: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.15% QD; Week 2; Test type: Superiority; p = 0.0009, MMRM; Difference in LS Mean = -25.12, 95% CI 2-sided [-39.84 to -10.41]
Statistical Analysis 2: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% BID; Week 2; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -47.85, 95% CI 2-sided [-62.64 to -33.06]
Statistical Analysis 3: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.5% QD; Week 2; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -41.04, 95% CI 2-sided [-56.00 to -26.08]
Statistical Analysis 4: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% QD; Week 2; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -45.05, 95% CI 2-sided [-59.69 to -30.40]
Statistical Analysis 5: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.15% QD; Week 2; Test type: Superiority; p = 0.1806, MMRM; Difference in LS Mean = 9.99, 95% CI 2-sided [-4.66 to 24.63]
Statistical Analysis 6: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.5% QD; Week 2; Test type: Superiority; p = 0.4333, MMRM; Difference in LS Mean = -5.93, 95% CI 2-sided [-20.82 to 8.95]
Statistical Analysis 7: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% QD; Week 2; Test type: Superiority; p = 0.1805, MMRM; Difference in LS Mean = -9.94, 95% CI 2-sided [-24.51 to 4.63]
Statistical Analysis 8: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% BID; Week 2; Test type: Superiority; p = 0.0895, MMRM; Difference in LS Mean = -12.74, 95% CI 2-sided [-27.45 to 1.98]
Statistical Analysis 9: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.15% QD; Week 8; Test type: Superiority; p = 0.0042, MMRM; Difference in LS Mean = -28.38, 95% CI 2-sided [-47.74 to -9.02]
Statistical Analysis 10: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 0.5% QD; Week 8; Test type: Superiority; p = 0.0003, MMRM; Difference in LS Mean = -36.52, 95% CI 2-sided [-56.03 to -17.01]
Statistical Analysis 11: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% QD; Week 8; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -45.19
Statistical Analysis 12: Comparison: DB: Vehicle BID vs DB: Ruxolitinib 1.5% BID; Week 8; Test type: Superiority; p < 0.0001, MMRM; Difference in LS Mean = -57.15, 95% CI 2-sided [-76.53 to -37.77]
Statistical Analysis 13: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.15% QD; Week 8; Test type: Superiority; p = 0.4243, MMRM; Difference in LS Mean = 7.78, 95% CI 2-sided [-11.37 to 26.93]
Statistical Analysis 14: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 0.5% QD; Week 8; Test type: Superiority; p = 0.9715, MMRM; Difference in LS Mean = -0.35, 95% CI 2-sided [-19.65 to 18.95]
Statistical Analysis 15: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% QD; Week 8; Test type: Superiority; p = 0.3507, MMRM; Difference in LS Mean = -9.03, 95% CI 2-sided [-28.05 to 9.99]
Statistical Analysis 16: Comparison: DB: TAC 0.1% BID/Vehicle Cream BID vs DB: Ruxolitinib 1.5% BID; Week 8; Test type: Superiority; p = 0.0320, MMRM; Difference in LS Mean = -20.98, 95% CI 2-sided [-40.15 to -1.82]

5. Secondary Outcome: Percentage of Participants Who Achieve a ≥ 50% Improvement From Baseline in EASI (EASI-50) at Weeks 2, 4, and 8
Description: The categorical variable EASI-50 will be equal to 1 for percentage improvement from baseline in EASI score of 50% or greater and will be equal to 0 for percentage improvement of less than 50%. This definition is introduced for the purpose of identifying participants who respond to the treatment (1 = responder, 0 = non-responder).
Time Frame: Week 2, 4 and 8
Population: ITT Population included all participants who are randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 52 | 50
percentage of participants
  Week 2 | 13.5 | 43.1 | 31.4 | 57.1 | 50.0 | 52.0
  Week 4 | 23.1 | 66.7 | 52.9 | 58.8 | 73.1 | 78.0
  Week 8 | 26.9 | 60.8 | 54.9 | 62.7 | 69.2 | 76.0

6. Secondary Outcome: Percentage Change From Baseline in EASI Score at Week 4
Description: as for outcome 1
Time Frame: Baseline and Week 4
Population: ITT Population included all participants who are randomized to the study. Overall number of participants analyzed are participants with data available for analysis at Week 4.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 44 | 46 | 47 | 47 | 49 | 49
percent change | -15.5 (65.71) | -59.8 (35.71) | -45.4 (53.96) | -52.2 (48.32) | -67.0 (26.28) | -71.6 (25.27)

7. Secondary Outcome: Time to Achieve EASI-50
Description: Time to EASI-50 is defined as the interval between the time of randomization and the time of achieving at least 50% improvement in EASI score.
Time Frame: From Baseline to Week 8
Population: ITT population included all participants who are randomized to the study.
Measure: Median (Full Range); unit: week
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 52 | 50
week | 4 [0 to 8] | 2 [0 to 8] | 4 [0 to 8] | 2 [0 to 8] | 2 [0 to 8] | 2 [0 to 8]

8. Secondary Outcome: Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 to 1 Who Have an Improvement of ≥ 2 Points From Baseline at Weeks 2, 4, and 8
Description: IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). An IGA responder was defined as a participant achieving an IGA score of 0 to 1 and an IGA score improvement at least 2 from baseline.
Time Frame: Week 2, 4 and 8
Population: ITT Population included all participants who are randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 52 | 50
percentage of participants
  Week 2 | 1.9 | 11.8 | 5.9 | 4.1 | 13.5 | 8.0
  Week 4 | 7.7 | 25.5 | 9.8 | 13.7 | 21.2 | 38.0
  Week 8 | 9.6 | 17.6 | 15.7 | 31.4 | 30.8 | 48.0

9. Secondary Outcome: Mean Change From Baseline in the Itch Numerical Rating Scale (NRS) Score at Weeks 2, 4, and 8
Description: The Itch NRS is a once-per-24 hours ("daily") participant-reported measure of itch intensity to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours. The categorical NRS is defined as 0 = None, 1 to 3 = Mild, 4 to 6 = Moderate, and 7 to 10 = Severe.
Time Frame: Baseline, Week 2, 4 and 8
Population: ITT Population included all participants who are randomized to the study. Overall number of participants analyzed are participants with data available for analysis at specified time-point and 'n' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- DB: TAC 0.1% BID/ Vehicle BID: Participants applied triamcinolone 0.1% cream BID for 4 weeks followed by vehicle cream for 4 weeks in DB period.
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/ Vehicle BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 48 | 44 | 46 | 48 | 48 | 47
score on scale
  Baseline | 6.0 (2.11) | 5.2 (2.22) | 6.1 (2.23) | 6.2 (1.71) | 6.2 (2.14) | 5.9 (2.25)
  Change from Baseline at Week 2: number analyzed (Participants) | 42 | 39 | 44 | 43 | 45 | 45
  Change from Baseline at Week 2 | -0.7 (1.46) | -2.2 (1.75) | -1.9 (1.97) | -2.5 (2.23) | -3.1 (2.14) | -3.7 (2.56)
  Change from Baseline at Week 4: number analyzed (Participants) | 37 | 38 | 41 | 40 | 44 | 45
  Change from Baseline at Week 4 | -1.0 (1.79) | -2.5 (1.94) | -2.3 (2.08) | -2.6 (2.22) | -3.3 (2.24) | -4.0 (2.89)
  Change from Baseline at Week 8: number analyzed (Participants) | 33 | 33 | 38 | 38 | 39 | 37
  Change from Baseline at Week 8 | -1.2 (2.13) | -2.2 (1.86) | -3.0 (2.49) | -2.9 (2.41) | -3.8 (2.39) | -4.2 (2.91)

10. Secondary Outcome: Number of Participants With At Least One Adverse Event (AEs) and as Per Severity
Description: AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. The severity of AEs was assessed using CTCAE v4.03 Grades 1 through 4.Data are reported for Grade 3 and higher severity for this outcome measure.
Time Frame: Up to Week 24
Population: Safety Population in the DB treatment period included all enrolled participants who applied at least 1 dose of ruxolitinib cream, triamcinolone cream, or vehicle cream.
Measure: Count of Participants; unit: Participants
Groups:
- OL: Vehicle BID to Ruxolitinib 1.5% BID; OL: TAC BID/Vehicle Cream BID to Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID; OL: Ruxolitinib 1.5% BID: Following DB Period, at Week 8, participants who met criteria (compliant with the protocol and no safety concerns) received open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks
Arm/Group | DB: Vehicle BID | DB: TAC 0.1% BID/Vehicle Cream BID | DB: Ruxolitinib 0.15% QD | DB: Ruxolitinib 0.5% QD | DB: Ruxolitinib 1.5% QD | DB: Ruxolitinib 1.5% BID | OL: Vehicle BID to Ruxolitinib 1.5% BID | OL: TAC BID/Vehicle Cream BID to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.15% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 0.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% QD to Ruxolitinib 1.5% BID | OL: Ruxolitinib 1.5% BID
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 51 | 50 | 41 | 40 | 45 | 41 | 42 | 43
Participants
  At Least One AE | 17 | 17 | 19 | 11 | 17 | 12 | 5 | 11 | 11 | 8 | 11 | 17
  Grade 3 and Higher | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 24
Groups:
- Vehicle BID: Participants applied vehicle cream BID for 8 weeks. At Week 8, participants who met criteria were offered open-label treatment with Ruxolitinib 1.5% cream BID for 4 weeks.
- Triamcinolone 0.1% BID for 4 Weeks Then 4 Week Vehicle BID: Participants applied triamcinolone 0.1% cream BID for 4 weeks followed by vehicle cream for 4 weeks. At Week 8, participants who met criteria were offered open-label treatment with ruxolitinib 1.5% cream BID for 4 weeks.
- INCB018424 0.15% QD: Participants applied Ruxolitinib 0.15% cream QD for 8 weeks. At Week 8, participants who met criteria were offered open-label treatment with Ruxolitinib 1.5% cream BID for 4 weeks.
- INCB018424 0.5% QD: Participants applied Ruxolitinib 0.5% cream QD for 8 weeks. At Week 8, participants who met criteria were offered open-label treatment with Ruxolitinib 1.5% cream BID for 4 weeks.
- INCB018424 1.5% QD: Participants applied Ruxolitinib 1.5% QD for 8 weeks. At Week 8, participants who met criteria were offered open-label treatment with Ruxolitinib 1.5% cream BID for 4 weeks.
- INCB018424 1.5% BID: Participants applied Ruxolitinib 1.5% cream BID for 8 weeks. At Week 8, participants who met criteria were offered open-label treatment with Ruxolitinib 1.5% cream BID for 4 weeks.
Arm/Group | Vehicle BID | Triamcinolone 0.1% BID for 4 Weeks Then 4 Week Vehicle BID | INCB018424 0.15% QD | INCB018424 0.5% QD | INCB018424 1.5% QD | INCB018424 1.5% BID
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/51 | 0/51 | 0/51 | 0/259
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/51 | 0/51 | 0/51 | 0/51 | 0/259
Other Adverse Events (participants affected / at risk) | 10/52 | 3/51 | 6/51 | 2/51 | 6/51 | 23/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle BID (N=52) | Triamcinolone 0.1% BID for 4 Weeks Then 4 Week Vehicle BID (N=51) | INCB018424 0.15% QD (N=51) | INCB018424 0.5% QD (N=51) | INCB018424 1.5% QD (N=51) | INCB018424 1.5% BID (N=259)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle BID (N=52) | Triamcinolone 0.1% BID for 4 Weeks Then 4 Week Vehicle BID (N=51) | INCB018424 0.15% QD (N=51) | INCB018424 0.5% QD (N=51) | INCB018424 1.5% QD (N=51) | INCB018424 1.5% BID (N=259)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 4 (6) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 13 (17)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT03011892/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03011892/SAP_001.pdf